CLINICAL TRIAL: NCT02702076
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of Continuous Subcutaneous Infusion in Parkinson's Disease Patients With Refractory Visual Hallucinations
Brief Title: Apomorphine in Parkinson's Disease Patients With Visual Hallucinations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Teus van Laar, MD PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL55949
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Parkinson's Disease; Hallucinations, Visual
Keywords: Apomorphine
MeSH Terms: conditions — Parkinson Disease; Hallucinations | interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apomorphine (Experimental): This arm will be treated with continuous subcutaneous infusion of apomorphine. The infusion will start with 1 mg/hr during the waking day (approximately 16 hours). The flow rate will be adjusted on a weekly basis, and may be increased with 0.5 to 1.0 mg/hr per discretion of the investigator, aiming at the disappearance of visual hallucinations. The duration of treatment is 4 weeks.
  Interventions: Drug: Apomorphine
- Placebo (Placebo Comparator): This arm will be treated with continuous subcutaneous infusion of placebo. The infusion will start with 1 mg/hr during the waking day (approximately 16 hours). The flow rate will be adjusted on a weekly basis, and may be increased with 0.5 to 1.0 mg/hr per discretion of the investigator aiming at the disappearance of visual hallucinations. The duration of treatment is 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apomorphine — Continuous subcutaneous infusion of apomorphine during waking day
  Other Names: APO-go; N04BC07
  Arms: Apomorphine
Drug: Placebo — Continuous subcutaneous infusion of placebo during waking day
  Arms: Placebo

SUMMARY:
This randomised, double-blind, placebo-controlled trial will evaluate the efficacy of continuous apomorphine infusion compared to placebo in PD patients with visual hallucinations, inadequately controlled with clozapine and cholinesterase inhibitors.

DETAILED DESCRIPTION:
Introduction Visual hallucinations occur frequently in Parkinson's disease (PD). The prevalence of visual hallucinations ranges from 22 to 38%, increasing after long-term follow-up to more than 60%. Risk factors for visual hallucinations are age, disease duration, and cognitive impairment. The treatment of visual hallucinations is cumbersome and options are limited. Only clozapine has been proven to be efficacious without deteriorating the motor symptoms of PD. Instead of oral dopamine agonists and rotigotine, continuous infusion of apomorphine is well-tolerated in PD patients with cognitive impairments and/or visual hallucinations. Even beneficial effect of apomorphine on visual hallucinations are suggested, however there is lack of a randomized controlled trial.

The purpose of this randomised, double-blind, placebo-controlled trial is to evaluate the efficacy of continuous apomorphine infusion compared to placebo in PD patients with visual hallucinations, inadequately controlled with clozapine and cholinesterase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged ≥30;
* Diagnosis of established PD, defined by the Movement Disorders Society PD criteria (Postuma et al., 2015);
* Presence of visual severe hallucinations defined as more than 3 times a week (van Laar et al., 2010);
* Visual hallucinations must have developed after PD diagnosis;
* Visual hallucinations must have been optimally treated with reduction of dopamine agonists if possible, and prescription of clozapine and/or cholinesterase inhibitors if needed;
* Female subjects must complaint with a highly effective contraceptive method (oral hormonal contraception alone is not considered highly effective and must be used in combination with a barrier method) during the study, if sexually active;
* Subjects should be able and capable of adhering to the protocol, visit schedules, and medication intake according to the judgement of the investigator.

Exclusion Criteria:

* Symptomatic, clinically relevant and medically uncontrolled orthostatic hypotension;
* Patients with a prolonged QT interval corrected for heart rate according to Bazett's formula (QTc) of >450 ms for male and >470 ms for female at screening, or history of a long QT syndrome;
* PD medication change (i.e., dopamine-agonists, amantadine, monoamine oxidase (MAO)-B inhibitors, anticholinergics and cholinesterase inhibitors) in last month prior to initiation (van Laar et al., 2010);
* Active psychosis or a history of significant psychosis;
* Any medical condition that is likely to interfere with an adequate participation in the study including e.g. current diagnosis of unstable epilepsy, clinically relevant cardiac dysfunction and/or myocardial infarction or stroke within the last 12 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression of Severity | Four weeks
  Clinical Global Impression of Severity questionnaire

SECONDARY OUTCOMES:
Clinical Global Impression of Improvement | Four weeks
  Clinical Global Impression of Improvement questionnaire
Cognition | Four weeks
  Montreal Cognitive Assessment
Depression | Four weeks
  Hamilton Anxiety and Depression Scale
Anxiety | Four weeks
  Hamilton Anxiety and Depression Scale
Motor symptoms | Four weeks
  Part III of Movement Disorders Society - Unified Parkinson's Disease Rating Scale
Motor complications | Four weeks
  Part IV of Movement Disorders Society - Unified Parkinson's Disease Rating Scale
Sleeping problems | Four weeks
  Parkinson's Disease Sleep Scale
Neuropsychiatric symptoms | Four weeks
  Neuropsychiatric Inventory - Questionnaire
Visual Hallucinations | Four weeks
  Dutch Visual Hallucinations Questionnaire
Attention | Four weeks
  Reaction Time Task
Visual perception | Four weeks
  Visual Object and Space Perception battery
Apathy | Four weeks
  Apathy Scale
Quality of Life | Four weeks
  Parkinson's Disease Questionnaire (shortened version)

OTHER OUTCOMES:
Blood pressure | Four weeks
  Orthostatic blood pressure measurement
Occurrence of adverse events | Four weeks
  Occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Teus van Laar, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Department of Neurology, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Laar T, Postma AG, Drent M. Continuous subcutaneous infusion of apomorphine can be used safely in patients with Parkinson's disease and pre-existing visual hallucinations. Parkinsonism Relat Disord. 2010 Jan;16(1):71-2. doi: 10.1016/j.parkreldis.2009.05.006. Epub 2009 Jun 12. No abstract available. PMID 19524477
- [Result] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Result] Fenelon G, Alves G. Epidemiology of psychosis in Parkinson's disease. J Neurol Sci. 2010 Feb 15;289(1-2):12-7. doi: 10.1016/j.jns.2009.08.014. Epub 2009 Sep 8. PMID 19740486
- [Result] Goetz CG, Ouyang B, Negron A, Stebbins GT. Hallucinations and sleep disorders in PD: ten-year prospective longitudinal study. Neurology. 2010 Nov 16;75(20):1773-9. doi: 10.1212/WNL.0b013e3181fd6158. Epub 2010 Oct 20. PMID 20962287
- [Result] Gallagher DA, Parkkinen L, O'Sullivan SS, Spratt A, Shah A, Davey CC, Bremner FD, Revesz T, Williams DR, Lees AJ, Schrag A. Testing an aetiological model of visual hallucinations in Parkinson's disease. Brain. 2011 Nov;134(Pt 11):3299-309. doi: 10.1093/brain/awr225. Epub 2011 Sep 15. PMID 21921019
- [Result] Borgemeester RW, Drent M, van Laar T. Motor and non-motor outcomes of continuous apomorphine infusion in 125 Parkinson's disease patients. Parkinsonism Relat Disord. 2016 Feb;23:17-22. doi: 10.1016/j.parkreldis.2015.11.013. Epub 2015 Nov 22. PMID 26709292
- [Result] Garcia Ruiz PJ, Sesar Ignacio A, Ares Pensado B, Castro Garcia A, Alonso Frech F, Alvarez Lopez M, Arbelo Gonzalez J, Baiges Octavio J, Burguera Hernandez JA, Calopa Garriga M, Campos Blanco D, Castano Garcia B, Carballo Cordero M, Chacon Pena J, Espino Ibanez A, Gorospe Onisalde A, Gimenez-Roldan S, Granes Ibanez P, Hernandez Vara J, Ibanez Alonso R, Jimenez Jimenez FJ, Krupinski J, Kulisevsky Bojarsky J, Legarda Ramirez I, Lezcano Garcia E, Martinez-Castrillo JC, Mateo Gonzalez D, Miquel Rodriguez F, Mir P, Munoz Fargas E, Obeso Inchausti J, Olivares Romero J, Olive Plana J, Otermin Vallejo P, Pascual Sedano B, Perez de Colosia Rama V, Perez Lopez-Fraile I, Planas Comes A, Puente Periz V, Rodriguez Oroz MC, Sevillano Garcia D, Solis Perez P, Suarez Munoz J, Vaamonde Gamo J, Valero Merino C, Valldeoriola Serra F, Velazquez Perez JM, Yanez Bana R, Zamarbide Capdepon I. Efficacy of long-term continuous subcutaneous apomorphine infusion in advanced Parkinson's disease with motor fluctuations: a multicenter study. Mov Disord. 2008 Jun 15;23(8):1130-6. doi: 10.1002/mds.22063. PMID 18442107
- [Result] Martinez-Martin P, Reddy P, Antonini A, Henriksen T, Katzenschlager R, Odin P, Todorova A, Naidu Y, Tluk S, Chandiramani C, Martin A, Chaudhuri KR. Chronic subcutaneous infusion therapy with apomorphine in advanced Parkinson's disease compared to conventional therapy: a real life study of non motor effect. J Parkinsons Dis. 2011;1(2):197-203. doi: 10.3233/JPD-2011-11037. PMID 23934921
- [Result] Martinez-Martin P, Reddy P, Katzenschlager R, Antonini A, Todorova A, Odin P, Henriksen T, Martin A, Calandrella D, Rizos A, Bryndum N, Glad A, Dafsari HS, Timmermann L, Ebersbach G, Kramberger MG, Samuel M, Wenzel K, Tomantschger V, Storch A, Reichmann H, Pirtosek Z, Trost M, Svenningsson P, Palhagen S, Volkmann J, Chaudhuri KR. EuroInf: a multicenter comparative observational study of apomorphine and levodopa infusion in Parkinson's disease. Mov Disord. 2015 Apr;30(4):510-6. doi: 10.1002/mds.26067. Epub 2014 Nov 10. PMID 25382161
- [Result] Ellis C, Lemmens G, Parkes JD, Abbott RJ, Pye IF, Leigh PN, Chaudhuri KR. Use of apomorphine in parkinsonian patients with neuropsychiatric complications to oral treatment. Parkinsonism Relat Disord. 1997 Apr;3(2):103-7. doi: 10.1016/s1353-8020(97)00009-6. PMID 18591063